CLINICAL TRIAL: NCT07307534
Title: Central Nevus Removal Versus Conservative Treatment for Halo Nevus With Vitiligo: A Prospective Randomized Controlled Trial
Brief Title: Nevus Removal vs. Conservative Treatment in Halo Nevus With Vitiligo: A Randomized Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJPF-LCY-V2025121
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Vitiligo; Halo Nevus
Keywords: Vitiligo; Halo nevus; Randomized Controlled Trial; Tacrolimus; NB-UVB; Nevus excision; Treatment comparison; Efficacy; Safety; VASI score
MeSH Terms: conditions — Vitiligo; Nevus, Halo

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized controlled study. Participants are randomly assigned to two groups, receiving central nevus excision plus medication or conservative medication only, respectively. The study aims to compare the efficacy and safety of the two interventions for treating halo nevus accompanied by non-segmental vitiligo.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Central Nevus Excision Group (Experimental): Participants in this arm undergo surgical or laser excision of the central nevus, with standardized medication initiated one week postoperatively.
  Interventions: Procedure: Central Nevus Excision; Combination Product: The Standardized Medication Regimen
- Conservative Treatment Group (Active Comparator): Participants in this arm receive standardized medication only without nevus removal.
  Interventions: Combination Product: The Standardized Medication Regimen

INTERVENTIONS:
Procedure: Central Nevus Excision — Participants undergo removal of the central halo nevus based on its diameter:
  Diameter <0.3 cm: CO₂ laser ablation. Diameter ≥0.3 cm: Surgical excision. All procedures are performed under local anesthesia with strict aseptic technique. Postoperative care and wound management are provided according to standard protocols.
  Arms: Central Nevus Excision Group
Combination Product: The Standardized Medication Regimen — For stable disease, apply topical 0.1% tacrolimus ointment twice daily combined with NB-UVB phototherapy once every other day.
  For active or progressive cases, oral prednisone (prednisone acetate, 0.3 mg/kg/day) is added to the above stable-stage regimen.

SUMMARY:
This clinical trial aims to compare the efficacy and safety of central nevus removal versus conservative treatment in patients with halo nevus accompanied by non-segmental vitiligo. It is a single-center, prospective, randomized controlled trial involving 60 participants aged 6 to 45 years, who will be randomly assigned to either the nevus removal group or the conservative treatment group. The removal group will undergo surgical or laser excision of the central nevus followed by medication, while the conservative group will receive medication only. Both groups will be followed for 6 months. Outcomes include repigmentation assessment using vitiligo scoring indices, quality of life measures, and serial serum cytokine profiling. The study seeks to provide high-level evidence to guide clinical management of halo nevus with vitiligo. Key points:

1. For patients with halo nevus accompanied by non-segmental vitiligo.
2. For patients aged 6 to 45 years.
3. Compares nevus excision and conservative treatment.
4. Follows participants for 6 months.
5. Focuses on effectiveness and safety.

DETAILED DESCRIPTION:
Background:

Halo nevus and vitiligo are both autoimmune pigment loss disorders that frequently co-occur and share overlapping immune pathways. Current management of halo nevus with vitiligo remains controversial: removal of the central nevus may eliminate an immune target and promote repigmentation but carries risks of Koebner phenomenon and scarring; conservative treatment avoids procedural trauma but may yield slower or suboptimal responses. Robust prospective comparisons of these strategies are lacking.

1. Study Design:

   Single-center, randomized controlled trial. Sixty patients with halo nevus and non-segmental vitiligo (BSA ≤2%) will be randomized 1:1 to the excision group or the conservative group.
2. Excision group: Central nevus removal via CO₂ laser (if diameter <0.3 cm) or surgical excision (if ≥0.3 cm), followed by standardized medication after 1 week.
3. Conservative group: Standardized medication only, without nevus removal. The standardized medication regimen is as follows:

   For stable disease, apply topical 0.1% tacrolimus ointment twice daily combined with NB-UVB phototherapy once every other day.

   For active or progressive cases, oral prednisone (prednisone acetate, 0.3 mg/kg/day) is added to the above stable-stage regimen.
4. Duration: 6 months with follow-ups at 1, 3, 6 months.
5. Outcome Measures:

   Primary Endpoint: Percentage of participants achieving VASl50 response Secondary Endpoints: Percentage of participants achieving VASI75 and VASI90 responses at each follow-up time point; changes in VASI, VSAS, VES, VETF scores; proportion of participants achieving lGA score improvement; patient-reported outcomes (DLQI/CDLQI, VitiQoL); incidence of treatment-emergent adverse events Other Pre-specified Outcomes: Changes in 12 serum cytokines (IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-17, IFN-α, IFN-γ, TNF-α).
6. Statistical Methods: Categorical data will be presented as frequencies and percentages, continuous data as mean ± SD. Between-group comparisons will use chi-square tests, Fisher's exact test, independent t-test, or Mann-Whitney U test as appropriate. Multivariate analysis will employ logistic regression. SPSS, R 4.3.2, and GraphPad Prism will be used for analysis (significance: p ≤ 0.05). The primary and secondary efficacy endpoints will be analyzed using the intention-to-treat (ITT) principle, with sensitivity analysis performed on the per-protocol (PP) population.
7. Ethics & Compliance: Approved by the Ethics Committee of the First Affiliated Hospital of Air Force Medical University. Informed consent is obtained from all participants' guardians.
8. Significance: This trial will systematically evaluate the clinical and immunological effects of central nevus removal versus conservative management in halo nevus with vitiligo, aiming to optimize treatment strategies and provide evidence-based guidance for clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with halo nevus accompanied by non-segmental vitiligo, with BSA ≤2% (excluding acral regions).

  * Central nevus confirmed as benign melanocytic nevus through clinical observation and dermatoscope.

    * Age 6 to 45 years, regardless of gender ④ Physically able to tolerate surgery and local anesthesia

Exclusion Criteria:

* History of keloid formation or hypertrophic scarring (to avoid abnormal hyperplasia at the operative site and interference with repigmentation assessment)

  * Other autoimmune diseases (e.g., hyperthyroidism)

    * Patients with significant endocrine disorders, psychiatric conditions, hematologic diseases, hepatic/renal disorders, cardiovascular/cerebrovascular diseases, severe infections, or other major systemic illnesses

      * Use of hormonal medications, immunomodulators, or phototherapy within the past 1 month ⑤ Pregnant or lactating women ⑥ Allergy to anesthetic agents or excipients

        * Poor psychological status or compliance, unable to cooperate with postoperative follow-up or care ⑧ Concurrent conditions requiring other treatments that may interfere with the study observations

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving VASl50 Response | From enrollment to the end of treatment at 6 months.
  VASl (Vitiligo Area and Severity lndex) 50 response is defined as a 50% or greater reduction in VASl score from baseline. Assessment is conducted by trained dermatologists using standardized VASl scoring criteria.

SECONDARY OUTCOMES:
Percentage of Participants Achieving VASI75 and VASI90 responses at each follow-up time point | From enrollment to the end of treatment at 6 months.
  VASl75 (or VASI90) response is defined as a 75% (or 90%) or greater reduction in VASl score from baseline. Assessment is conducted by trained dermatologists using standardized VASl scoring criteria.
Change in Vitiligo Area and Severity Index (VASl) Score | From enrollment to the end of treatment at 6 months.
  Calculate the difference between the VASl score at 6 months and the baseline VASl score, including the mean percentage change in VASI from baseline at 6 months. This reflects the improvement vitiligo area and severity over the treatment period.
Change in Vitiligo Signs of Activity Score (VSAS) Score | From enrollment to the end of treatment at 6 months.
  Calculate the difference between the VSAS score at 6 months and the baseline VSAS score.
Change in Vitiligo Extent Score (VES) Score | From enrollment to the end of treatment at 6 months.
  Calculate the difference between the VES score at 6 months and the baseline VES score.
Change in Vitiligo European Task Force (VETF) Score | From enrollment to the end of treatment at 6 months.
  Calculate the difference between the VETF score at 6 months and the baseline VETF score.
Change in Dermatology life quality index (DLQI) Score | From enrollment to the end of treatment at 6 months.
  Description & Structure: Dermatology Life Quality Index (DLQI) is a 10-item, disease-specific quality of life questionnaire designed for adults with skin conditions. It assesses the impact of skin disease across three domains: Physical, Social, and Psychological impacts. Children Dermatology life quality index (CDLQI) is the children's version of the DLQI, which is suitable for children aged 5 to 16 years. For young children, parental assistance or proxy completion is recommended.
  Scoring Range: Each item is rated on a 4-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Quite a lot", 3 = "Very much"). The total score is the sum of all 10 items, ranging from 0 to 30.
  Score Direction & Interpretation: A higher total score indicates a greater negative impact on the child's disease-specific quality of life (a worse outcome). A decrease in the score from baseline represents an improvement in quality of life.
Change in The Vitiligo-specific Quality-of-Life instrument (VitiQoL) Score | From enrollment to the end of treatment at 6 months.
  Description & Structure: The VitiQoL is a 15-item, disease-specific quality of life questionnaire designed for patients with vitiligo. It comprises three subdomains: Psychological Burden, Activity Limitation, and Appearance Concerns. Patients are asked to recall their experience over the past week and rate how bothered they have been by each item on a 5-point Likert scale (0 = "Never", 1 = "Rarely", 2 = "Sometimes", 3 = "Often", 4 = "Always").
  Scoring Range: The total score ranges from 0 to 60, calculated by summing the scores of all 15 items.
  Score Direction & Interpretation: A higher total score indicates greater impairment in disease-specific quality of life (worse outcome). A decrease in score from baseline represents an improvement.
Proportion of Participants Achieving investigator Global Assessment (lGA) Score lmprovement | From enrollment to the end of treatment at 6 months.
  Assess participants' lGA scores at 24 weeks. Participants with an lGA score of "mild" or better (score s 2) are defined as achieving improvement, and the proportion is calculated.
Incidence of Treatment-Emergent Adverse Events | From enrollment to the end of treatment at 6 months.
  All surgery-related and disease-related adverse events, such as localized erythema, pruritus, scarring, and Koebner phenomenon, will be documented and analyzed, including their incidence, severity, and association with the interventions.

OTHER OUTCOMES:
Changes in levels of 12 serum cytokines | From enrollment to the end of treatment at 6 months.
  Venous blood will be collected from the elbow at baseline and at 1, 3, and 6 months post-treatment to measure 12 serum cytokines (IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-17, IFN-α, IFN-γ, TNF-α). The changes in levels will be statistically analyzed to explore their correlation with clinical response and the underlying mechanisms of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Jian, Principal Investigator — First Affiliated Hospital of Air Force Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No